CLINICAL TRIAL: NCT05774093
Title: Evaluation of COVID-19 Immune Barrier and Reinfection Risk
Acronym: COVID
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Bingliang, Principal Investigator, Sun Yat-sen University
Other Study IDs: COVID-19 Immune Barrier Study
Record Dates: First submitted 2023-03-12; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: COVID-19 Infection; Immunization; Infection
MeSH Terms: conditions — COVID-19; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1.peripheral blood sample;2.COVID-19 nucleic acid specimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Antibody Group 1: Participants will be divided into positive group and negative group according to the baseline of COVID-19 antibody titer.Group 1 is for those COVID-19 antibody are positive.
- COVID-19 Antibody Group 2: Participants will be divided into positive group and negative group according to the baseline of COVID-19 antibody titer.Group 1 is for those COVID-19 antibody are negative.

SUMMARY:
The goal of this observational study is to evaluate the protective effect of immune barrier on secondary infection after COVID-19 (coronavirus disease 2019) vaccination or COVID-19 virus Omicron B A. 5.2 strain infection by dynamically monitoring the COVID-19 antibody titer, cellular immune function and the occurrence of secondary infection of healthy participants, mainly medical staff in our hospital, to understand the cross protective effect of COVID-19 antibody on different variants of Omicron, and explore the best time to use COVID-19 vaccine to strengthen immunity after Omicron mutant infection.

DETAILED DESCRIPTION:
This study is a single center, prospective, non-intervention study. It is planned to recruit 300 medical and nursing participants, administrative and logistics participants or other participants who can cooperate with the follow-up for 48 weeks to voluntarily join the group.

Participants will be investigated about the vaccination history of COVID-19 vaccine, whether they have ever been infected with COVID-19, the time of initial infection with COVID-19, and following clinical symptoms.The COVID-19 antibody titer of peripheral blood will be used for baseline.

The participants will be divided into positive group and negative group according to the COVID-19 antibody titer results,then they wii be followed up for 48 weeks.If the participants have no symptoms related to COVID-19 infection, COVID-19 antibody and COVID-19 nucleic acid will be tested every 4-8 weeks according to the epidemic situation (the specific visit time is initially set as 0 week, 6 ± 2 weeks, 12 ± 4 weeks, 20 ± 4 weeks, 28 ± 4 weeks, 36 ± 4 weeks, 48 ± 4 weeks). There will be about 7 visits in total, according to the epidemic situation and the time of secondary infection of the participants). If the nucleic acid turns to be positive, we will consider it as the asymptomatic infection, then we will collect nasal/pharyngeal swabs for gene sequencing of virus strains, and terminate the study.

If the participants get fever, fatigue, sore throat, cough, nasal congestion, runny nose, muscle soreness or headache and other symptoms related to COVID-19 infection during the study period, they need to test the COVID-19 antigen or COVID-19 nucleic acid within 48 hours. If it is positive, we will collect nasal/pharyngeal swabs for gene sequencing of virus strains, and terminate the study in advance.

ELIGIBILITY:
Inclusion Criteria:

1. No age limit, no gender limit;
2. Medical staff, administrative and logistics staff who work in the Third Affiliated Hospital of Sun Yat-Sen University or other participants who can cooperate with the follow-up for 48 weeks;
3. The participants need to be sure whether they have ever been infected with COVID-19, and need to be clearly remember the time when they first infected with COVID-19.

Exclusion Criteria:

1. Have the following serious respiratory diseases: such as asthma, bronchiectasis, chronic obstructive pulmonary disease, pulmonary interstitial disease, tuberculosis and other respiratory diseases that may interfere with symptom observation;
2. Those with other serious diseases or disease history that affect immune function, including but not limited to uncontrolled and unresectable malignant tumors,hematological diseases, cachexia, active bleeding, severe malnutrition, mental diseases, autoimmune diseases, HIV, etc.
3. Those who have long-term assignment plans and cannot return to the hospital regularly for follow-up.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The participants need to be sure whether they have ever been infected with COVID-19, and need to be clearly remember the time when they first infected with COVID-19.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of COVID-19 reinfection in COVID-19 antibody positive and negative groups. | 48weeks
  This study is an observational study. The incidence of COVID-19 reinfection is mainly based on the participants with positive COVID-19 nucleic acid test. The proportion of participants with positive COVID-19 nucleic acid test in the total number during the observation period after 48 weeks observation will be counted.

SECONDARY OUTCOMES:
Dynamic changes of COVID-19 antibody titer in 48 weeks after COVID-19 infection. | 48weeks
  We will test COVID-19 antibody every 4-8 weeks and record the data to observe the dynamic change of titer.
Dynamic changes of cellular immune function in 48 weeks after COVID-19 infection. | 48weeks
  Flow cytometry will be used to detect the cellular immune function of participants every 4-8 weeks, and record data to analyze its dynamic changes.
Antibody titer of COVID-19 in uninfected persons. | 48weeks
  The "uninfected person" refers to the participant who is still uninfected with COVID-19 at the end of our study. We will record and analyze the dynamic change of COVID-19 antibody titer within 48 weeks.
The cellular immune function of COVID-19 in uninfected persons. | 48weeks
  We will record and analyze the dynamic change of the cellular immune function by flow-cytometry within 48 weeks.
The change of antibody titer in uninfected people after COVID-19 vaccine. | 48weeks
  We will test and analyze the changes of COVID-19 antibody titer of uninfected people within 48 weeks after the booster immunization with COVID-19 vaccine.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Hall VJ, Foulkes S, Charlett A, Atti A, Monk EJM, Simmons R, Wellington E, Cole MJ, Saei A, Oguti B, Munro K, Wallace S, Kirwan PD, Shrotri M, Vusirikala A, Rokadiya S, Kall M, Zambon M, Ramsay M, Brooks T, Brown CS, Chand MA, Hopkins S; SIREN Study Group. SARS-CoV-2 infection rates of antibody-positive compared with antibody-negative health-care workers in England: a large, multicentre, prospective cohort study (SIREN). Lancet. 2021 Apr 17;397(10283):1459-1469. doi: 10.1016/S0140-6736(21)00675-9. Epub 2021 Apr 9. PMID 33844963
- [Result] Michlmayr D, Hansen CH, Gubbels SM, Valentiner-Branth P, Bager P, Obel N, Drewes B, Moller CH, Moller FT, Legarth R, Molbak K, Ethelberg S. Observed protection against SARS-CoV-2 reinfection following a primary infection: A Danish cohort study among unvaccinated using two years of nationwide PCR-test data. Lancet Reg Health Eur. 2022 Sep;20:100452. doi: 10.1016/j.lanepe.2022.100452. Epub 2022 Jun 30. PMID 35791335
- [Result] Servellita V, Syed AM, Morris MK, Brazer N, Saldhi P, Garcia-Knight M, Sreekumar B, Khalid MM, Ciling A, Chen PY, Kumar GR, Gliwa AS, Nguyen J, Sotomayor-Gonzalez A, Zhang Y, Frias E, Prostko J, Hackett J Jr, Andino R, Wadford DA, Hanson C, Doudna J, Ott M, Chiu CY. Neutralizing immunity in vaccine breakthrough infections from the SARS-CoV-2 Omicron and Delta variants. Cell. 2022 Apr 28;185(9):1539-1548.e5. doi: 10.1016/j.cell.2022.03.019. Epub 2022 Mar 18. PMID 35429436